CLINICAL TRIAL: NCT03396211
Title: An Open-Labeled, Phase I Study to Evaluate the Safety and Tolerability of Apatinib With Nivolumab in Patients With Unresectable or Metastatic Cancer
Brief Title: A Study to Evaluate Apatinib (Also Known as Rivoceranib) Plus Nivolumab in Participants With Unresectable or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSK-AM107
Record Dates: First submitted 2017-12-21; First posted 2018-01-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Cancer
Keywords: Metastatic; Unresectable
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — apatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apatinib with Nivolumab (Experimental): Participants will receive an oral dose of apatinib once per day with a fixed dose of nivolumab given intravenously every 2 weeks.
  Interventions: Drug: Apatinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Apatinib — Apatinib tablets
  Other Names: Rivoceranib, Apatinib Mesylate
Drug: Nivolumab — Fixed dose of nivolumab given intravenously every 2 weeks
  Other Names: Opdivo

SUMMARY:
This is an open-labeled, single-center, Phase I study to evaluate the safety, tolerability, and efficacy of apatinib with nivolumab treatment in participants with unresectable or metastatic cancer. Total study duration will be approximately 50 months: 12 months of recruitment plus 6 months of treatment and subsequent survival follow up.

DETAILED DESCRIPTION:
Primary objectives:

* To evaluate the safety and tolerability of apatinib with nivolumab in participants with unresectable or metastatic cancer.
* To assess efficacy by objective response rate (ORR), best overall response (BOR), time to response (TTR), and duration of response (DoR) per response evaluation criteria for solid tumors (RECIST) v1.1 and/or response evaluation criteria for solid tumors for immune-based therapeutics (iRECIST).
* To assess disease control rate (DCR), and duration of disease control (DDC) by RECIST v1.1, and/or iRECIST.

Secondary objectives:

* To evaluate the efficacy of apatinib with nivolumab in participants with unresectable or metastatic cancer as measured by:
* Overall survival (OS)
* Progression-free survival (PFS)
* Event-free survival (EFS)

ELIGIBILITY:
Inclusion Criteria:

1. Documented primary diagnosis of histologic- or cytologic-confirmed solid tumor cancer inclusive of gastric adenocarcinoma, renal cell carcinoma, melanoma, non-small cell lung cancer (NSCLC), breast cancer, angiosarcoma, leiomyosarcoma, synovial sarcoma, and alveolar soft part sarcoma or other solid tumor for which anti-Vascular endothelial growth factor receptor (VEGFR)2 targeted therapy could be applicable.
2. Locally advanced unresectable or metastatic disease.
3. Nivolumab treatment naive and able to begin nivolumab treatment concurrently with initiation of apatinib or have received at least 3 doses of nivolumab treatment and are continuing nivolumab therapy.
4. 1 or more measurable lesions per RECIST v1.1.
5. Participants who have adequate bone-marrow, renal and liver function including:

   1. Hematologic: absolute neutrophil count ≥ 1,500/ cubic millimetre (mm^3), platelets≥ 100,000/mm^3, hemoglobin ≥ 9.0 grams (g)/ per decilitre (dL) (blood transfusion to meet the inclusion criteria within 2 weeks is not allowed).
   2. Renal: serum creatinine < 1.5× upper limit of normal (ULN); urinary protein should be< 2+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥ 2+, then a 24-hour urine or urine protein/creatinine ratio must be collected and must demonstrate <2 g of protein in 24 hours to allow participation in the study.
   3. Hepatic: serum bilirubin < 1.5× ULN, aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0× ULN(≤ 4.0× ULN, if with liver metastases).
   4. Blood coagulation tests: Partial thromboplastin time (PTT) and international normalized ratio (INR) ≤ 1.5× ULN and ≤ 1.5×ULN, respectively.
6. Eastern Cooperative Oncology Group (ECOG) performance status are evaluated to be ≤ 1 (Participants with ECOG performance status of 2 may be enrolled only with advance review and written approval by the medical monitor).
7. Expected survival of ≥ 12 weeks, in the judgement of the investigator.
8. Ability to swallow the study drug tablets.

Exclusion Criteria:

1. History of another malignancy within 2 years prior to enrollment, unless it does not pose a significant risk to life expectancy as per the investigator.
2. Central nervous system (CNS) metastases as shown by radiology records or clinical evidence of symptomatic CNS involvement in the last 3 months prior to enrollment. Participants are eligible if metastases have been treated and have returned to neurologic baseline or are neurologically stable (except for residual signs or symptoms related to the CNS treatment).
3. Cytotoxic chemotherapy, surgery, radiotherapy or other targeted therapies and checkpoint inhibitors (excluding nivolumab if not nivolumab treatment naive) within 3 weeks (4 weeks in cases of ramucirumab, mitomycin C, nitrosourea, lomustine; 1 week in case of biopsy) prior to enrollment (adjuvant radiotherapy given to local area for non-curative symptom relief is allowed until 2 weeks before enrollment).
4. Any other therapies including biological and approved therapies within 3 half-lives or 3 weeks whichever is longer and have not recovered from all toxicities from the treatment.
5. Therapy with clinically significant systemic anticoagulant or anti thrombotic agents within 7 days prior to enrollment that may prevent blood clotting and, in the investigator's opinion, could place the participants at risk. Maximum dose of 325 milligram (mg)/day of aspirin is allowed.
6. History of bleeding diathesis or clinically significant bleeding within 14 days prior to enrollment.
7. History of clinically significant thrombosis (bleeding or clotting disorder) within the past 3 months prior to enrollment that, in the investigator's opinion, may place the participant at risk of side effects from anti-angiogenesis products.
8. History of gastrointestinal bleeding, gastric stress ulcerations, or peptic ulcer disease within the past 3 months prior to enrollment that, in the investigator's opinion, may place the participant at risk of side effects from anti-angiogenesis products.
9. Myocardial infarction or an unstable angina pectoris within 3 months prior to enrollment.
10. Prior major surgery or fracture within 3 weeks prior to enrollment or presence of any non-healing wound (procedures such as catheter placement are not considered to be major).
11. Participation in any other interventional clinical trial, within 4 weeks prior to enrollment or while participating in this study.
12. Previous treatment with apatinib.
13. Hypersensitivity to apatinib or components of its formulation.
14. History of uncontrolled hypertension ([HTN], blood pressure ≥ 140/90 millimeters of mercury [mmHg]) and change in anti hypertensive medication within 7 days prior to enrollment) that is not well managed by medication and the risk of which may be precipitated by VEGF inhibitor therapy.
15. History of severe adverse events including uncontrolled HTN or other common anti-angiogenesis class drug effects that were related to ramucirumab or bevacizumab discontinuation and/or may indicate a higher risk to the safety of the participant if provided further anti-angiogenesis treatment, in the investigator's opinion.
16. History of symptomatic congestive heart failure (New York Heart Association III-IV), symptomatic or poorly controlled cardiac arrhythmia, complete left bundle branch block, bifascicular block, or any clinically significant ST segment and/or T-wave abnormalities, QTcF>450 msec for males or QTcF > 470 msec for females prior to enrollment.
17. Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9, and CYP2C19.
18. History of drug or alcohol abuse within past 5 years.
19. Known history of human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS).
20. Known history of positive tests for hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.
21. Pregnant or breast-feeding females.
22. Active bacterial infections.
23. Presence of substance abuse, medical, psychological, or social illness(es)that, in the judgement of the investigator, may interfere with the participant's participation or safety, or which may impact the objectives of the study.
24. History of clinically significant glomerulonephritis, biopsy-proven tubulointerstitial nephritis, crystal nephropathy, or other renal insufficiencies.
25. Gastrointestinal malabsorption, or any other condition that in the opinion of the investigator might affect the absorption of the study drug.
26. Grade 2 or greater toxicity from ongoing nivolumab treatment and irAE including colitis and pneumonitis, if not nivolumab treatment naive.
27. Active autoimmune disease or a history of known autoimmune disease.
28. History of drug-induced interstitial pneumonitis or severe hypersensitivity to other antibody therapies.
29. Known or underlying medical condition (for example, a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would make the administration of study drug hazardous to the participant or obscure the interpretation of toxicity determination or adverse events.
30. Other conditions that, in the judgement of the investigator, contraindicate study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to approximately 5 years
Objective Response Rate (ORR): Percentage of Participants who Achieve Confirmed Complete Response (CR) or Partial Response (PR) | Up to approximately 5 years
  ORR per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and/or iRECIST criteria.
Best Overall Response Rate (BOR) | Up to approximately 5 years
  BOR is the best response, according to RECIST v1.1 and/or RECIST criteria, recorded over the duration of the study until disease progression, or recurrence.
Time To Response (TTR) | Up to approximately 5 years
  TTR is the time lapsed from enrollment until documented response according to RECIST v1.1 and/or iRECIST criteria.
Duration of Response (DoR) | Up to approximately 5 years
  DoR is the time from documented tumor response (PR or CR) until disease progression or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 5 years
  DCR is the proportion of participants with radiologically documented stable or decreased tumor burden per RECIST v1.1 and/or iRECIST criteria.
Duration of Disease Control (DDC) | Up to approximately 5 years
  DDC is the time from enrollment until disease progression or death from any cause, whichever occurs first. Disease progression will be evaluated by RECIST v1.1 and/or iRECIST criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  OS is the time from participant enrollment until death from any cause.
Event Free Survival (EFS) | Up to approximately 5 years
  EFS is defined as time from enrollment to a > 20% increase tumor size from baseline by RECIST v1.1, development of distant metastatic disease, or death.
Progression Free Survival (PFS) | Up to approximately 5 years
  PFS is the time from start of apatinib treatment to either radiological progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States